CLINICAL TRIAL: NCT06918756
Title: The Development and Validation of a Cough Control Questionnaire
Brief Title: Development of a Cough Control Questionnaire (CCQ)
Acronym: CCQ
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH24-072
Record Dates: First submitted 2025-04-01; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cough
Keywords: patient-reported outcomes; cough; control; questionnaire
MeSH Terms: conditions — Cough | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Focus group cohort: Patients aged 18-100 with chronic cough including refractory chronic cough and unexplained chronic cough. Exclusions include: current smokers, ACE inhibitor use. Patients will be recruited to form focus groups to inform the creation of a cough control questionnaire. This will take the form of semi-structured interviews with open to closed questions. This same cohort will also engage in cognitive interviews after the preliminary cough control questionnaire has been made, to ensure that the language and wording is clear and appropriate. Recruitment will continue until thematic saturation is achieved.
  Interventions: Other: Focus group interviews
- Validation study cohort: Patients aged 18-100 with chronic cough will be recruited. Exclusion criteria include: current smokers, smoking within the last 12 months, use of angiotensin converting enzyme inhibitor (ACEi), respiratory tract infection within the last 4 weeks and limited English.
  Prospective consecutive patients with chronic cough will complete Cough Control Questionnaire, cough severity assessments and health status assessments. Patients will be invited to undergo objective cough frequency monitoring and cough challenge testing.

INTERVENTIONS:
Other: Questionnaires — Completion of new questionnaire in addition to other patient reported outcome measures that measure cough severity and cough-related quality of life.
Other: Focus group interviews — Semi-structured focus group interviews for patients with refractory chronic cough
  Groups: Focus group cohort
Other: Objective cough measures — Cough monitoring and cough sensitivity testing.

SUMMARY:
Chronic cough (>8 weeks in duration) affects 5-12% of the global population, and is associated with considerable health status impairment and comorbidities. Currently, there are validated severity and impact outcome measures whilst objective measures with cough frequency monitoring is not available in routine clinical practice. Unlike other chronic respiratory diseases, namely asthma, there are no validated dedicated tools to assess the control of cough as a disease.

This study aims to develop a validated patient-focused tool to assess the control of cough, which may be useful to evaluate the benefit and value of treatments in both clinical and research settings.

DETAILED DESCRIPTION:
This study will involve 3 phases:

* Phase 1: Literature review. Review of currently available validated tools to assess control in respiratory diseases.
* Phase 2: Development of Cough Control Questionnaire (CCQ). Patient focus groups will aid development of a conceptual framework of cough control and ensure content validity through qualitative research methods including thematic analysis. Expert panel review of cough control framework will also be undertaken. CCQ item development will be grounded in patient focus groups and expert review findings, and reviewed through cognitive debrief with patients.
* Phase 3: Validation of CCQ. Prospective consecutive patients with chronic cough will complete CCQ, cough severity assessments and health status assessments. Patients will be invited to undergo objective cough frequency monitoring and cough challenge testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 and over with acute and chronic cough (including refractory chronic cough and unexplained chronic cough) and able to read and write in English. A smaller number (n =20) of healthy volunteers will also be included with no evidence of significant respiratory disease.

Exclusion Criteria:

* Current smokers (or smoking within the last 12 months), respiratory tract infection within the last 4 weeks, use of angiotensin converting enzyme inhibitors (ACEi), and pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients will be recruited from tertiary chronic cough clinics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
A questionnaire to assess cough control | 2 weeks
  The primary aim of the study is to develop and validate a cough control questionnaire which accurately reflects the nature of cough control.

SECONDARY OUTCOMES:
Cough severity | 2 weeks
  Assessed using dedicated patient reported outcome measures. Correlations with CCQ will be assessed.
Cough-related quality of life and health status | 2 weeks
  Assessed using dedicated patient reported outcome measures. Correlations with CCQ will be assessed.
Cough frequency | 2 weeks
  Cough frequency (Coughs/24 hours) will be assessed at visits using cough monitors and correlations with CCQ will be assessed.
Cough reflex testing | 2 weeks
  Capsaicin concentration for C2 and C5 (to elicit 2, and 5 coughs respectively) will be assessed in a subset of patients. Correlations with CCQ will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
As the project progresses, other sites may be added. Only pseudonymised data would be sent to other researchers, for the purpose of statistical analysis and results.